CLINICAL TRIAL: NCT04440995
Title: The Effects of Perioperative PECS Block on Postoperative Pain Control During Robotic Breast Surgery and Breast Reconstruction - Double Blind Randomized Controlled Trial -
Brief Title: The Effects of Perioperative PECS Block During Robotic Breast Surgery and Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2020-0430
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Breast Neoplasm
Keywords: breast neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS block(P) group (Experimental): PECS group (P) received general anesthesia and pectoral nerve block(PECS block) with 025% ropivacaine after surgical resection of breast by operator.
  Interventions: Procedure: pectoral nerve block
- Control(c) group (No Intervention): only received general anesthesia

INTERVENTIONS:
Procedure: pectoral nerve block — Patients received standardized general anesthesia. PECS block were applied under vision using blunted tip cannula(27G, 30mm) after surgical resection of breast by operator. 0.25% ropivacaine 10ml was injected into fascia between pectoralis major and minor muscles. 0.25% ropivacaine 20ml was injected into fascia between pectoralis minor and serratus anterior muscles at the level of the third rib. Breast reconstruction is performed after PECS block
  Arms: PECS block(P) group

SUMMARY:
Pectoral nerve blocks (PECS blok) are used in postoperative analgesia after breast surgery in nowadays. Many studies shows that pectoral nerve blocks is effective for reducing pain and postoperative opioid consumption undergoing mastectomy. This study was planned to evaluate the efficacy of intraoperative PECS block for postoperative analgesia after robot breast surgery and immediate breast reconstruction.

DETAILED DESCRIPTION:
Sixty patients were randomly allocated into two groups by computerised process, each including 30 patients. PECS group (P) received general anesthesia and pectoral nerve block(PECS block) with 025% ropivacaine after surgical resection of breast by operator. Control group(C) only received general anesthesia.

A Patient -controlled analgesia(PCA) device provides fentanyl for postoperative pain control.

The Primary outcome measures total dose of fentanyl consumption during the postoperative 24 hours, and secondary outcome measures pain scores at rest and movement.

ELIGIBILITY:
Inclusion Criteria:

1. 20years or older
2. Scheduled for robot-assisted nipple-sparing mastectomy with immediate gel implant or tissue expander breast reconstruction
3. American Society of Anesthesiologists(ASA) physical status I and III

Exclusion Criteria:

1. Emergency operation
2. Reoperation
3. Patients with local anesthetic allergy
4. Patients with coagulopathy
5. Patients on anticoagulants
6. Patients who cannot use patient controlled analgesia(PCA)
7. Patients with morbid obesity [body mass index (BMI) >35 kg/m2]
8. Patients with history of uncontrolled hypertension (diastolic BP >110mmHg) or DM
9. Patients with history of heart failure (unstable angina, congestive heart failure)
10. Patients with history of liver failure, renal failure, allergic to medicine
11. Patients with history of cerebrovascular disease (cerebral hemorrhage, cerebral ischemia)
12. Patients with history of uncontrolled psychiatric disease (PTSD, anxiety, depression)
13. Patients who cannot read the consent form (examples: Illiterate, foreigner)
14. Patients who withdraw the consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Total dose of fentanyl consumption during the postoperative 24h | after 24 hours postoperative period
  To evaluate the effect of PECS block undergoing robot-assisted nipple-sparing mastectomy (RANSM) with immediate breast reconstruction (IBR), total cumulative dose of fentanyl was measured for the first postoperative 24h

SECONDARY OUTCOMES:
a numeric rating score at rest | 0 hour after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 0.5 hour after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 1 hour after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 2 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 4 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 6 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 8 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 12 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at rest | 24 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 0 hour after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 0.5 hour after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 1 hour after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 2 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 4 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 6 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 8 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 12 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)
a numeric rating score at movement | 24 hours after surgery
  Secondary outcome measures were postoperative pain using numeric rating score (NRS, 0-10; 0=no pain and 10=worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jun Bai, Ph.D, Study Director — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No